CLINICAL TRIAL: NCT01105416
Title: Emergency Department Based Prevention Intervention to Delay Alcohol Use by Young Adolescents
Brief Title: Emergency Department (ED) Adolescent Alcohol Prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, James Linakis Ph.D., Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0088-08; R21AA018380 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Alcohol Drinking
Keywords: Pediatric Emergency Department; Parental monitoring; Adolescent; Parents; Communication; Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Standard Care (ESC) (Placebo Comparator): Standard emergency department care plus informational brochures
  Interventions: Behavioral: ESC
- Brief Prevention Intervention (BPI) (Experimental): Brief Prevention Intervention in the Pediatric ED
  Interventions: Behavioral: Brief Prevention Intervention (BPI)

INTERVENTIONS:
Behavioral: Brief Prevention Intervention (BPI) — Brief Prevention Intervention: Participants will receive the BPI, a brief, family-focused prevention intervention in the Pediatric ED. The session will be comprised of parent-targeted skill building directed primarily at parental monitoring and the importance of parent-adolescent communication as the precursor to successful monitoring.
  Arms: Brief Prevention Intervention (BPI)
Behavioral: ESC — Enhanced standard care
  Arms: Enhanced Standard Care (ESC)

SUMMARY:
The aim of the present study is to prevent or delay the initiation of alcohol use among young adolescents being seen in a pediatric emergency department, by enhancing parental monitoring and improving parent/adolescent conversations. Previous studies have shown that the pediatric emergency department is an excellent location for performing prevention interventions. By targeting individuals and their families in the pediatric emergency department (PED), we are capitalizing on the opportunity to perform a prevention intervention among a high risk population when parent and youth may be particularly receptive to the intervention.

DETAILED DESCRIPTION:
Our long term goal is to develop, implement, and evaluate a program to prevent or delay the initiation of alcohol use in young adolescents by increasing protective factors and reducing risk through a family-based brief prevention intervention started in the pediatric emergency department (PED). The primary aims of the proposed developmental study include: (1) To pilot test a prevention intervention in alcohol-naïve adolescents, make necessary revisions, and finalize an intervention manual and (2) conduct a randomized pilot trial comparing the prevention intervention with enhanced standard care. After conducting an open trial of the prevention intervention with 10 adolescents, ages 12-14, and their accompanying parent(s), and refining the intervention, we will use a two-group randomized design to test the hypothesis that the prevention intervention will prevent/delay the initiation of alcohol use significantly more than enhanced standard care only. 100 adolescents, ages 12-14, who present to the PED and their accompanying parent(s)/caregiver will be enrolled into the study. Eligible, assenting adolescents and their consenting parent(s)/caregiver will complete a series of assessment instruments relating to alcohol and other drug (AOD) use, communication styles, parenting styles, and alcohol attitudes and behaviors. Parent/youth family units will then be randomly assigned to one of two conditions: 1) Enhanced Standard Care (ESC) or 2) Brief Targeted Prevention Intervention with Boosters (BTP). The initial session will be comprised of parent-targeted skill building directed primarily at parental monitoring and the importance of parent-adolescent communication as the precursor to successful monitoring. The primary goal of the prevention session will be the mobilization of the parents' own resources to increase communication and monitoring using motivational interviewing techniques. Parents within this condition will also receive periodic brochures and telephone booster sessions at 1 and 3 months to explore parental implementation of the plan from the previous session(s) and make revisions as necessary. Adolescents and parents will then be reassessed six months following their PED visit. Adolescents will also be assessed with monthly, brief, web-based follow-up contacts to determine the status of their alcohol use.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents, age 12-14, who are being seen in the Pediatric ED for a non life-threatening injury and their parent/caregiver;
2. Adolescent must be medically stable;
3. For a parent/adolescent family unit to be eligible, one or both of the adolescent's parents must be present in the ED with the adolescent; and
4. The adolescent must report not having initiated alcohol use.

Exclusion Criteria:

1. Family units in which either the parent or the adolescent are cognitively unable to take part in the intervention;
2. Those in which the youth is suspected by the clinical staff of being a victim of child abuse (these adolescents will be reported to child protective services);
3. Those in which the youth is medically or surgically unstable;
4. Family units in which the adolescent is being evaluated for a possible psychiatric disorder; and those without a telephone and/or a verifiable address of residence.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Parental monitoring | 2 years
  A one-tailed, α = 0.05 level of significance will be used to tests the difference between the BPI and ESC groups on hypotheses 2A on parental monitoring (using the PMQ and Parent/student self-check), 2B using the PMPI, drug use promoting peers, and parent/child beliefs and peers, 2C using scales on parent attitudes and parent beliefs about drug use, and 2D using intentions to use scale from the CTC.

CONTACTS AND LOCATIONS:
Overall Officials: James G Linakis, PhD, MD, Principal Investigator — University Emergency Medicine Foundation
Locations (1):
- Hasbro Children's Hospital Emergency Department, Providence, Rhode Island, United States